CLINICAL TRIAL: NCT02853214
Title: Identification of Genetic Factors Predisposing to Dysglobulinemia
Brief Title: Familial Dysglobulinemia
Acronym: PreFamDys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2007-460; 2007-A00644-49 (Other: ID-RCB)
Record Dates: First submitted 2016-07-13; First posted 2016-08-02 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Dysglobulinemia
Keywords: Dysglobulinemia; Multiple Myeloma; MGUS; Waldenström; genetic factors; Sequencing
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Identification of genetic factors in dysglobulinemia cases (Experimental)
  Interventions: Genetic: Genetic analysis of peripheral blood samples

INTERVENTIONS:
Genetic: Genetic analysis of peripheral blood samples — M.D investigators report the identified families with all the information: description of the familial area (for example: 2 cases father and son), last medical report for the case with the type of dysglobulinemia, monoclonal component isotype, medical background and contact information for one of the patients or cases with Name/surname/Date of Birth/address and phone. They contact the patient to explain the study and establish the family pedigree. They collect the information on all the family members and send to the patient a mail: an information note on the study, a prescription for the blood sample and the informed consents. They proceed in the same way for the relatives with the additional prescription: EIP. They organize the logistic in the medical lab or hospital chosen by the person. They receive 4 Heparin and 1 serum tubes for each and with this, they obtain a large amount of biological material for the genetic analysis thanks to the establishment of lymphoblastoid cell lines

SUMMARY:
Multiple Myeloma (MM) is a malignant proliferation of monoclonal plasma cells. Myeloma accounts for almost 14% of all hematologic cancers and is essentially incurable. Myeloma commonly evolves from a precursor disease, Monoclonal gammopathy of undetermined significance (MGUS). Despite intensive study, the etiology of MGUS and myeloma are unknown and no lifestyle or environmental exposure factors have been identified that are consistently linked to increased risk of MM, MGUS or the transition between the two.

The overall goal is to identify risk genes for dysglobulinemia, and more specifically Multiple Myeloma. This will involve the conservation of cells in a bank and genetic sequencing on samples obtained from families with at least two cases of dysglobulinemia. Material used for sequencing is likely to include fresh peripheral blood cells or lymphoblastoid lines established from peripheral blood lymphocytes of patients.

ELIGIBILITY:
Inclusion Criteria:

* 2 cases per family at least
* 1 case alive at least
* biological material available for 1 case at least
* Patients give their informed consent
* attached to the French Health protection service

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1868 (Actual)
Dates: Start 2008-02-06 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Data of a bank cells, clinically annotated, from families with at least 2 cases of dysglobulinemia and at least 1 case alive.plasma cell dysplasia | up to 48 months
  The investigator collects blood samples from patients with dysglobulinemia and their relatives and with this, the investigators constitutes the bank cells thanks to the establishment of lymphoblastoid cell lines.
  The investigator considers as "dysglobulinemia" cases patients with Multiple Myeloma, MGUS, Waldenström's disease and MGUS (monoclonal gammopathy of unknown significance ) as wells as plasmacytomas confirmed histologically or cytologically.

SECONDARY OUTCOMES:
Single Nucleotide Polymorphism array for identification of polymorphisms predictive of dysglobulinemia | at day 0
  The biological material, obtained from fresh peripheral blood cells and from Lymphoblastoid cells lines, is used for pangenic sequencing. It allows to better understand the mechanism of genetic variations who could be involve in the myeloma genesis

CONTACTS AND LOCATIONS:
Overall Officials: Charles DUMONTET, Principal Investigator — Hospices Civils de Lyon
Locations (47):
- France (47):
  - Service d'Oncologie-Radiothérapie - CHU Pointe-à-Pitre/Abymes Guadeloupe, Pointe à Pitre, Guadeloupe
  - Service de Médecine Interne-Hématologie, CHU de Fort de France Fort de France, Fort-de-France, Martinique
  - CHU d'ABBEVILLE, Abbeville
  - CHU Amiens Picardie, Amiens
  - CHU Groupe Hospitalier Sud Hématologie Clinique, Amiens
  - CH d'Avignon, Avignon
  - CHU de Besançon, Besançon
  - CH de Blois Service d'Hématologie, Blois
  - Hôpital Avicenne Service d'Hématologie, Bobigny
  - Service d'Hématologie clinique et Thérapie Cellulaire, CHU de BORDEAUX, Bordeaux
  - CHU Morvan, Brest
  - Service d'hématologie Clinique, Caen
  - Hématolgie- Hôpital privé Cesson-Sévigné, Cesson-Sévigné
  - CH William Morey, Service d'Hémato-Oncologie, Chalon-sur-Saône
  - CHU de Chartres, Chartres
  - Département d'Oncogénitique - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Sud Francilien, Corbeil-Essonnes
  - Service d'Hématologie Clinique, CHU de Dijon, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - GHM, Institut Daniel Hollard, Grenoble
  - CHU Albert Michallon, Grenoble
  - Service d'Hématologie, CHU de Versailles, Le Chesnay
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans
  - Service d'Onco-hématologie, Hôpital Saint-Vincent GH-ICL, Lille
  - Service des Maladies du Sang CHU Lille, Lille
  - Département d'Oncogénétique, Centre Paoli Calmettes, Marseille
  - CHR-Metz-Thionville, Hôpital de Mercy, Service d'Hématologie, Metz
  - CHU d'Annecy, Metz-Tessy
  - Hôpital Saint-Eloi, Département d'Hématologie clinique, Montpellier
  - Service d'Oncologie Médical, Centre Azuréen de Canrérologie-1, Mougins
  - CHU-HÔTEL -Dieu de Nantes, Nantes
  - Hôpital de l'Archet 1, Nice
  - CHU Carémeau, Nîmes
  - Institut Curie, Paris
  - Hôpital St Antoine Service des maladies du Sang, Paris
  - Jean Paul FermandService Immuno-Hématologie Hôpital Saint Louis, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Hôpital Robert Debré Service du Professeur A. DELMER Hématologie Clinique, Reims
  - CHU de Rennes Hôpital Sud, Rennes
  - CH de Rodez, Rodez
  - Hôpital de Saint- Germain en Laye, Saint-Germain-en-Laye
  - Département d'Hématologie à l'Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Hôpital Purpan Service d'Hématologie, Toulouse
  - Centre Hospitalier de Valence, Valence
  - CHU de Nancy, Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumontet C, Demangel D, Galia P, Karlin L, Roche L, Fauvernier M, Golfier C, Laude MC, Leleu X, Rodon P, Roussel M, Azais I, Doyen C, Slama B, Manier S, Decaux O, Pertesi M, Beaumont M, Caillot D, Boyle EM, Cliquennois M, Cony-Makhoul P, Doncker AV, Dorvaux V, Petillon MO, Fontan J, Hivert B, Leduc I, Leyronnas C, Macro M, Maigre M, Mariette C, Mineur P, Rigaudeau S, Royer B, Vincent L, Mckay J, Perrial E, Garderet L. Clinical characteristics and outcome of 318 families with familial monoclonal gammopathy: A multicenter Intergroupe Francophone du Myelome study. Am J Hematol. 2023 Feb;98(2):264-271. doi: 10.1002/ajh.26785. Epub 2023 Jan 1. PMID 36588407